CLINICAL TRIAL: NCT05581628
Title: EVALUATION OF THE FREQUENCY OF FIBROMYALGIA IN PATIENTS WITH CELIAC DISEASE
Brief Title: FREQUENCY OF FIBROMYALGIA IN PATIENTS WITH CELIAC DISEASE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Okan Küçükakkas, Assoc. Prof., Bezmialem Vakif University
Other Study IDs: Bezmialem4494
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Celiac Disease; Fibromyalgia
MeSH Terms: conditions — Celiac Disease; Fibromyalgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Celiac Patients Group: Patients previously diagnosed with celiac disease by the gastroenterology clinic.
  Interventions: Diagnostic Test: Pain location inventory (PLI); Diagnostic Test: Symptom Impact Questionnaire (SIQR); Diagnostic Test: Fibromyalgia Impact Questionnaire (FIQ)

INTERVENTIONS:
Diagnostic Test: Pain location inventory (PLI) — PLI is obtained by questioning the pain in 28 regions in the last 7 days. Total score is between 0-28
Diagnostic Test: Symptom Impact Questionnaire (SIQR) — The SIQR score includes a total of 10 different evaluations in the last 7 days, including pain, energy, stiffness, sleep, depression, memory problems, anxiety, sensitivity to touch, balance problems, sensitivity to loud sounds-bright light-smells-cold. Each item is scored between 0-10 and the total score is obtained between 0-100. This total score is divided by 2 to get the SIQR score
Diagnostic Test: Fibromyalgia Impact Questionnaire (FIQ) — FIQ measures 10 different features, including physical function, well-being, absenteeism, difficulty at work, pain, fatigue, morning fatigue, stiffness, anxiety and depression. With the exception of the well-being trait, low scores indicate recovery or less affliction. The maximum possible score of each sub-title is 10. Thus, the total maximum score is 100.

SUMMARY:
950 / 5.000 Çeviri sonuçları Celiac disease is an autoimmune proximal small bowel disease that develops as a persistent intolerance to gluten-like gluten in cereals, mainly wheat gluten and other cereal proteins such as barley, rye, and oats in genetically susceptible individuals. Fibromyalgia syndrome (FMS) is a chronic musculoskeletal disease characterized by chronic widespread body pain, fatigue, morning stiffness, subjective swelling, sleep disturbance, intestinal problems, multiple somatic and cognitive problems, especially in the back, neck, shoulders and hips. In terms of intestinal symptoms, very similar findings can be observed between celiac disease and fibromyalgia. For this reason, the presence of celiac disease in FMS patients has been investigated in many studies and its frequency has been found to be high. However, the frequency of FMS in patients with celiac disease is not clear, and an overlooked diagnosis of fibromyalgia may leave many symptoms untreated.

ELIGIBILITY:
Inclusion Criteria:

Patients who agreed to participate in the study, signed the informed consent form, had the cognitive capacity to fill in the questionnaires and scales, and were followed up with a diagnosis of celiac will be included.

Exclusion Criteria:

Patients whose celiac diagnosis is uncertain, who do not agree to participate in the study, and who do not have sufficient cognitive capacity will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Statistical analysis of the demographic data of 60 patients diagnosed with celiac according to the ESPGHAN diagnostic criteria will be performed, and the frequency of comorbid diseases will be measured. The correlation between celiac disease and fibromyalgia will be determined and possible relationships between the two diseases will be investigated. The relationship between the presence and severity of fibromyalgia and celiac disease clinical types and modified marsh classification will be examined.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
Frequency of fibromyalgia | 3 months
  The frequency of fibromyalgia in celiac patients will be determined as percent.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No